CLINICAL TRIAL: NCT01547936
Title: A Single-Center Study Evaluating the Effect of the Controlled Adverse Environment (CAE) on Tear Film Stability Using the OPI 2.0 System, Ocular Protection Index (OPI), Tear Film Break-Up Time (TFBUT) and Mean Break up Area by Region (MBA) in Patients Diagnosed With Dry Eye Evaluated During Their Natural Blink Pattern
Brief Title: Effect of Controlled Adverse Environment (CAE) on Tear Film Stability
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-270-0002
Record Dates: First submitted 2012-02-15; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effect of the controlled adverse environment (CAE) on Mean Break-Up Area in subjects diagnosed with Dry Eye Syndrome.

DETAILED DESCRIPTION:
Single-Center, Pilot, controlled adverse environment (CAE) Study.

This is a single-center, one visit, pilot, CAE study. Dry Eye Subjects (N=30) who qualify will undergo tear film video recording, fluorescein staining, and break up time before CAE exposure and after CAE exposure.

All subjects will undergo baseline dry eye assessments including fluorescein staining, breakup time, conjunctival redness and tear film video recording. Subjects who qualify will then undergo CAE exposure for 90 minutes. At the end of CAE exposure subjects will undergo dry eye assessments again.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & either sex, any race
* Willing and able to follow all instructions
* Positive history of dry eye disease
* Use or desire to use drops for dry eye within the past 6 months

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy or lactating
* Use of disallowed medications
* Have ocular infections, or ocular conditions that could affect study parameters
* Have used an investigational drug or device within 30 days of start of study
* Female that is currently pregnant, planning a pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with dry eye disease
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change in tear film break up area | change from baseline in tear film break up area at 30 minutes post-CAE at study visit

SECONDARY OUTCOMES:
change in Fluorescein Staining | change from baseline in staining at 30 minutes post-CAE
Change in Tear film break up time (TFBUT) | change from baseline in tear film break up time at 30 minutes post-CAE
Change in Conjunctival Redness | change from baseline in conjunctival redness at 30 minutes post-CAE

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shazly, MD, Principal Investigator — Ophthalmic society of Egypt, Egyptian Glaucoma Society, American Acadamy of Ophthalmology, American Glaucoma Society, The association for research in vision and ophthalmology, international society of refractive surgery, Pan Arab Glaucoma Society
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States